CLINICAL TRIAL: NCT06178068
Title: Comparison of Bronchodilator Treatment Practices in Group E COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bugra Kerget, Associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/122
Record Dates: First submitted 2023-12-02; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: COPD Exacerbation Acute

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1; jet nebulizer group (Active Comparator): The Respirox® RNEB-18 device was used for the bronchodilator treatment given before the randomization of the patients and for the maintenance bronchodilator treatment given in Group 1 patients. After calibrating the device, it was determined that it performed nebulization with a flow of 6 lt/min.
  Interventions: Device: Comparison of bronchodilator effectiveness of nebulizer therapy devices
- Group 2; dry air nebulizer group (Active Comparator): In Group 2 patients, a HAVELSAN® EHSİM brand nebulizer produced in our country, compatible with the central system of our hospital, was used as a dry air nebulizer.
  Interventions: Device: Comparison of bronchodilator effectiveness of nebulizer therapy devices
- Group 3; Classic nebülizer group (Active Comparator): For classical nebulizer treatment in Group 3 patients, a nebulizer device compatible with our hospital's central oxygen system was used.
  Interventions: Device: Comparison of bronchodilator effectiveness of nebulizer therapy devices

INTERVENTIONS:
Device: Comparison of bronchodilator effectiveness of nebulizer therapy devices — The Respirox® RNEB-18 device was used for the bronchodilator treatment given before the randomization of the patients and for the maintenance bronchodilator treatment given in Group 1 patients. After calibrating the device, it was determined that it performed nebulization with a flow of 6 lt/min. In Group 2 patients, a HAVELSAN® EHSİM brand nebulizer produced in our country, compatible with the central system of our hospital, was used as a dry air nebulizer. For classical nebulizer treatment in Group 3 patients, a nebulizer device compatible with our hospital's central oxygen system was used. In Group 2 and 3 patients, the flow system could be adjusted manually. To be consistent with Group 1 patients, bronchodilator treatment was administered at a 6 lt/min flow rate.

SUMMARY:
COPD is a heterogeneous condition caused by airway (bronchitis/bronchiolitis) or alveolar (emphysema) abnormality, changes with chronic respiratory changes (dyspnea, dyspnoea, phlegm). It is characterized by persistent and frequently progressive airway obstruction. In COPD, which progresses with high mortality, non-pharmacological treatments are applied, as well as pharmacological treatments. They have an essential place in slowing down the progressive course of this treatment. However, despite the treatment administered to COPD patients, outdoor weather conditions, improper use of inhaler treatments, or comorbidities may cause acute exacerbation of COPD.

Dry air nebulizer devices use dry air from the central system in hospitals. This system, which converts bronchodilator drugs into nebulizers by creating high currents, works like classical nebulizers without an electrical system and can have a higher flow rate than jet nebulizer devices. This procedure, which can be applied to COPD patients without giving high-flow oxygen, prevents carbon dioxide retention. There is no study in the literature comparing the bronchodilator effectiveness of dry air, classical nebulizer, and jet nebulizer, and the investigators aimed to compare the efficacy of these three treatment modalities in our study.

ELIGIBILITY:
Inclusion Criteria:

* Group E COPD patients

Exclusion Criteria:

* Recent MI
* Pulmonary embolism
* Cerebral aneurysm
* Active hemoptysis
* Pneumothorax
* Nausea, vomiting
* Recent thorax, abdominal, and eye surgery were identified in the patients before the pulmonary function test and were not included in the study.
* Mental retardation
* Pneumonia with acute exacerbation of COPD
* Patients with pulmonary edema due to congestive heart failure
* Patients with interstitial lung disease along with COPD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the change in respiratory function test parameters after 5 days of nebulizer treatment applications.randomization on respiratory function tests | 5 days
  Measurement of % change in FVC, FEV1, RV, TLC level
Evaluation of the change in arterial blood gas parameters after 5 days of nebulizer treatment applications.randomization on respiratory function tests | 5 days
  Saturation %, measurement of change in partial oxygen and partial carbon dioxide levels in mm_Hg